CLINICAL TRIAL: NCT05368623
Title: Validation Study of RETINA-AI Galaxy™ v2.0, an Automated Diabetic Retinopathy Screening Device
Status: Completed | Type: Observational
Sponsor: RETINA-AI Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RETINA-AI-CT2
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetic Retinopathy; Diabetic Macular Edema; Diabetic Eye Problems
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Tomography, Optical Coherence; Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Sequential Enrollment: Patients aged 22yrs or older who have diabetes will be recruited from primary care settings.
  Interventions: Diagnostic Test: Color fundus photograph; Diagnostic Test: Optical Coherence Tomography (OCT) of the retina; Drug: Mydriatic Agent

INTERVENTIONS:
Diagnostic Test: Color fundus photograph — Subjects will undergo color fundus photography before and after pharmacological dilation of pupils.
Diagnostic Test: Optical Coherence Tomography (OCT) of the retina — Subjects will undergo OCT of the retina after pharmacological dilation of pupils.
Drug: Mydriatic Agent — Pharmacological dilation of pupils will be done by instilling mydriatic agent in eyes of Subjects

SUMMARY:
Diabetes affects over 37 million Americans and over 530 million people globally. Each diabetic patient needs at least one retinal exam per year starting immediately at the time of diagnosis if they have Type II diabetes (and starting at 5th year after disease onset if they have Type I diabetes). However, majority of diabetic patients do not get their eye exam due to multiple prohibitive factors such as cost, transportation, difficulty of taking time off from work, and inconvenience, amongst others. As a result, diabetes is the most common cause of visual impairment and blindness in working age adults in the United States and globally. Early detection via effective screening can prevent diabetes-related blindness. However, there are multiple barriers to screening. This prompted the development of RETINA-AI Galaxy™ v2.0, an automated Software as a Medical Device that screens for diabetic retinopathy in the primary care setting. This observational study was designed to validate the safety and efficacy of the RETINA-AI Galaxy™ Software-as-a-Medical-Device.

DETAILED DESCRIPTION:
This study was a prospective, multicenter, observational study to assess the safety and efficacy of the RETINA-AI Galaxy™ v2.0 ("Galaxy™") in screening for diabetic retinopathy in the primary care setting. The study design conformed to an Intent to Screen (ITS) paradigm. The Galaxy™ is a Software-as-a-Medical-Device designed to analyze digital color fundus photographs and rapidly screen for diabetic retinopathy in the primary care setting.

Subjects who met eligibility criteria were recruited from Sites in the United States staffed by primary care providers. Eligibility was assessed and informed consent was obtained, after which digital color fundus photographs were taken using U.S. Food and Drug Administration (FDA) cleared non-mydriatic fundus cameras, by an operator using the Galaxy photography manual.

There were a total of 3 non-mydriatic robotic screening cameras used in the AI system protocol part of the study. There was a dedicated validation camera used in the Validation Reading Center Protocol part of the study at each Site. Primary care clinical staff (e.g. medical assistant) with no prior professional ophthalmic photography experience and only a 4 hour training operated the RETINA-AI Galaxy v2.0 device and the screening cameras. The Retina Reading Center (RRC)- certified professional ophthalmic photographers operated the validation fundus cameras according the the 4W-D stereo protocol, and obtained OCT images of the macula.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patient age 22 or above
2. Patient with a documented diagnosis of diabetes as defined by any of the following:

   A. Hemoglobin A1c (HbA1c) ≥ 6.5% based on repeated assessments B. Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) based on repeated assessments C. Oral Glucose Tolerance test with 2-hour plasma glucose ≥ 200 mg/dL (11.1mmol/L) using equivalent of 75g anhydrous glucose dose in water.

   D. Symptoms of hyperglycemia or hyperglycemic crisis with random plasma glucose ≥ 200mg/dL (11.1 mmol/L) E. Criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA).
3. Understanding of the Study and willingness and ability to sign informed consent

EXCLUSION CRITERIA:

1. Persistent vision loss in one or both eyes
2. Diagnosis with macular edema, severe non-proliferative diabetic retinopathy, proliferative diabetic retinopathy, radiation retinopathy, or retinal vein occlusion.
3. History of retinal laser treatment, or injections into either eye, or any history of retinal surgery.
4. Currently enrolled in another interventional study of an investigational device or drug and actively receiving an investigational product for diabetic retinopathy (DR) or Diabetic Macula Edema (DME).
5. Subject has contraindication to mydriatic agent (dilating drops) or is unwilling or unable to dilate.
6. Subject is contraindicated from fundus photography (e.g. subject is hypersensitive to light).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects from Primary Care clinics - sampling method: non-probability, invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of RETINA-AI Galaxy v2.0 for diabetic retinopathy screening in the primary care setting. | 1 visit (1 day)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Research Organization, Los Angeles, California
  - Clinical Research Organization, Chicago, Illinois
  - Clinical Research Organization, Houston, Texas